CLINICAL TRIAL: NCT07307625
Title: A Randomized Comparative Study of Opioid-Free Versus Opioid-Based Anesthesia in Laparoscopic Cholecystectomy Surgery
Brief Title: LAPOFAR Trial: Opioid-Free vs. Remifentanil Anesthesia in Laparoscopic Cholecystectomy
Acronym: LAPOFAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gorkem Tukenmez, Resident Physician, Department of Anesthesiology and Reanimation, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DrLutfiKirdarTRH-ANES-GT-01; 2024/010.99/10/31 (Other: Ethics Approval Number)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management; Postoperative Nausea and Vomiting; Laparoscopic Cholecystectomy; Opioid-free Anesthesia; General Anesthesia
Keywords: Dexmedetomidine; Lidocaine; Opioid-Free Anesthesia; Analgesic Requirement; Postoperative Pain
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Lidocaine; Dexmedetomidine; Remifentanil

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel intervention groups. One group received opioid-free anesthesia (lidocaine and dexmedetomidine infusion), while the other received standard opioid-based anesthesia (remifentanil). Each participant remained in their assigned group throughout the procedure and follow-up period. The study used a 1:1 allocation ratio and compared outcomes such as postoperative pain, nausea and vomiting, and recovery parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-Free Anesthesia (OFA) (Experimental): Participants in this group received intravenous lidocaine and dexmedetomidine for opioid-free anesthesia. Lidocaine was administered as a 1.5 mg/kg bolus followed by a continuous infusion of 1.5 mg/kg/h. Dexmedetomidine was administered as a 0.5 µg/kg loading dose over 10 minutes, followed by an infusion of 0.5 µg/kg/h. No opioids were used intraoperatively. Standard induction with propofol and muscle relaxation with rocuronium were applied.
  Interventions: Drug: Lidocaine + Dexmedetomidine
- Opioid-Based Anesthesia (RA) (Active Comparator): Participants in this group received standard general anesthesia with remifentanil infusion at 0.1-0.5 µg/kg/min. Anesthesia induction was performed using propofol and rocuronium. All other surgical and anesthetic parameters were standardized to match those of the OFA group.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Lidocaine + Dexmedetomidine — Participants received intravenous lidocaine and dexmedetomidine as part of the opioid-free anesthesia protocol. Lidocaine was administered as a 1.5 mg/kg bolus followed by continuous infusion at 1.5 mg/kg/h. Dexmedetomidine was administered as a 0.5 µg/kg loading dose over 10 minutes, followed by continuous infusion at 0.5 µg/kg/h until the end of surgery. No intraoperative opioids were given.
  Arms: Opioid-Free Anesthesia (OFA)
Drug: Remifentanil — Participants received standard opioid-based anesthesia with continuous intravenous remifentanil infusion at 0.1-0.5 µg/kg/min. Induction and maintenance of anesthesia were standardized with propofol and rocuronium. All other perioperative conditions were matched to the OFA group.
  Arms: Opioid-Based Anesthesia (RA)

SUMMARY:
This study was a single-center, prospective, randomized clinical trial designed to compare the effects of opioid-free anesthesia (OFA) with standard opioid-based anesthesia during elective laparoscopic cholecystectomy. The aim was to evaluate the impact of these two anesthetic approaches on postoperative pain, analgesic requirement, hemodynamic stability, postoperative nausea and vomiting (PONV), and recovery quality.

A total of 101 patients, aged 18 to 65 years and classified as ASA I-II, undergoing elective laparoscopic cholecystectomy were enrolled and randomized into two groups. The OFA group received intravenous lidocaine and dexmedetomidine, while the standard anesthesia (RA) group received a remifentanil-based protocol. All other anesthetic agents and surgical procedures were standardized across both groups.

Intraoperative monitoring included heart rate, systolic and diastolic blood pressure, and end-tidal CO₂, recorded at 5-minute intervals. Postoperative assessments included visual analog scale (VAS) pain scores at multiple time points (10, 20, 30, 60 minutes; 2, 12, and 24 hours), rescue analgesic use, incidence of PONV, and Modified Aldrete Scores at 0, 30, and 60 minutes.

The results demonstrated that patients in the OFA group experienced significantly lower VAS pain scores in both early and late postoperative periods. The OFA group also required less rescue analgesia, had lower heart rate and blood pressure readings postoperatively, and showed a reduced incidence of PONV. Additionally, recovery parameters such as shorter time to extubation and higher early Aldrete scores favored the OFA group.

These findings suggest that opioid-free anesthesia using lidocaine and dexmedetomidine is a safe and effective alternative to opioid-based anesthesia in laparoscopic cholecystectomy. It provides better postoperative pain control, reduces opioid-related side effects, and improves overall recovery. The study supports the potential for integrating OFA into enhanced recovery protocols and calls for further multicenter trials with larger sample sizes to validate and generalize the results.

DETAILED DESCRIPTION:
Postoperative pain remains a major clinical concern, affecting recovery, patient comfort, and hospital resource utilization. Traditionally, opioids have played a central role in intraoperative and postoperative pain management. However, opioid use is associated with several adverse effects such as respiratory depression, nausea, vomiting, sedation, ileus, tolerance, hyperalgesia, and dependency. These drawbacks have driven interest in alternative strategies that reduce or eliminate perioperative opioid exposure, particularly within the framework of Enhanced Recovery After Surgery (ERAS) protocols.

Opioid-Free Anesthesia (OFA) is a multimodal approach that omits opioids and instead utilizes a combination of non-opioid agents such as lidocaine, dexmedetomidine, ketamine, NSAIDs, and magnesium sulfate to provide analgesia, hemodynamic stability, and sedation. OFA aims to minimize opioid-related side effects while maintaining effective pain control and facilitating faster recovery.

This single-center, prospective, randomized controlled trial was designed to compare OFA using intravenous lidocaine and dexmedetomidine to standard general anesthesia with remifentanil in patients undergoing elective laparoscopic cholecystectomy. The primary aim was to assess the effect of OFA on postoperative pain scores and rescue analgesia requirement. Secondary outcomes included intraoperative hemodynamic parameters, postoperative nausea and vomiting (PONV), and recovery quality assessed via Modified Aldrete Scores.

A total of 101 adult patients, aged 18-65 years, classified as ASA I-II, were enrolled and randomized into two groups:

OFA Group: Received intravenous lidocaine (1.5 mg/kg bolus followed by infusion at 1.5 mg/kg/h) and dexmedetomidine (0.5 μg/kg loading dose followed by 0.5 μg/kg/h infusion).

RA Group (Remifentanil Group): Received standard anesthesia with remifentanil infusion (0.1-0.5 μg/kg/min), in combination with propofol and rocuronium.

Standard monitoring included non-invasive blood pressure, ECG, SpO₂, EtCO₂, and bispectral index (BIS). Intraoperative hemodynamic values (heart rate, systolic and diastolic blood pressure, EtCO₂) were recorded at 5-minute intervals. Postoperative pain was assessed using the Visual Analog Scale (VAS) at 10, 20, 30, and 60 minutes, and at 2, 12, and 24 hours. PONV incidence and the need for rescue antiemetics were also recorded. Recovery was evaluated using Modified Aldrete Scores at 0, 30, and 60 minutes post-extubation.

Statistical analysis was performed using R (v4.5.1). Normality was assessed via the Shapiro-Wilk test. Between-group comparisons used the independent t-test or Mann-Whitney U test for continuous variables and chi-square or Fisher's exact test for categorical data. Within-group comparisons of pre- and postoperative values used paired t-tests or Wilcoxon signed-rank tests as appropriate.

The study found that the OFA group had significantly lower postoperative VAS scores at all time points, reduced need for rescue analgesics, and lower incidence of PONV. Hemodynamic parameters such as heart rate and blood pressure were more stable intra- and postoperatively in the OFA group. Moreover, time to extubation was shorter and early recovery scores were higher among patients who received OFA.

These findings suggest that opioid-free anesthesia with lidocaine and dexmedetomidine provides superior outcomes in terms of postoperative pain control, recovery, and complication rates compared to opioid-based anesthesia with remifentanil. The results support the inclusion of OFA in clinical practice and ERAS protocols for laparoscopic cholecystectomy. Further multicenter studies with larger sample sizes and inclusion of different surgical procedures are warranted to generalize these findings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* ASA I-II
* Elective laparoscopic cholecystectomy
* Informed consent
* BMI 18-30 kg/m²
* Normal liver and renal function

Exclusion Criteria:

* Refusal to participate
* Allergy to study drugs
* Chronic opioid use
* Major organ disease
* Pregnancy or lactation
* Open surgery conversion
* Recent participation in another trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score (VAS) | 0-24 hrs
  VAS at multiple time points post-surgery

SECONDARY OUTCOMES:
Rescue Analgesic Use | 0-24 hrs
  Total mg of analgesics
PONV Incidence | 0-24 hrs
  Presence of nausea/vomiting
Hemodynamic Monitoring | Intraoperative
  HR, SBP, DBP every 5 min
Recovery Score (Aldrete) | 0, 30, 60 min post-extubation
  Modified Aldrete score
Extubation Time | Immediately after surgery
  Minutes to extubation

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared publicly due to local data privacy regulations and institutional policy. Aggregate results will be available in published form.